CLINICAL TRIAL: NCT04070859
Title: Evaluation of Internal Fixation Of Glenoid Fractures
Brief Title: Fixation of Glenoid Fractures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Diaa El-Din Mohamed, Assistant Lecturer, Assiut University
Other Study IDs: Glenoid Fractures Fixation
Record Dates: First submitted 2019-07-21; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Glenoid; Fracture
Keywords: internal fixation
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Internal Fixation of Glenoid Fractures — Internal Fixation via (Paltes & Screws, Tension bands. etc)

SUMMARY:
Scapula fractures are uncommon but make up 3-5% of all shoulder girdle injuries. Moreover, intraarticular glenoid fossa fractures represent only 1% of scapula fractures.

They are frequently found with concomitant injuries to chest, head, brachial plexus and humerus.

The glenoid is an oval shaped portion on the lateral border of the scapula that articulates with the circular rounded end of the humeral head.

Superiorly the glenoid is part of the superior shoulder suspensory complex (SSSC) consisting of superior glenoid, coracoid process, coracoclavicular ligaments, distal end of the clavicle, acromioclavicular joint, coracoacromial ligament and acromial process.

Subsequently, stability of the shoulder is a complex mechanism in which muscles, ligamentous and capsular restraints, the labrum and joint vacuum, each play a role depending on position and activity.

The history of patients with glenoid fractures will mostly consist of either shoulder dislocation or direct trauma to the humeral head. The affected arm is "pseudo-paralysed" and supported in adduction and internal rotation.

Because of a thick layer of soft tissue, only mild swelling and ecchymosis may be seen .

For the diagnosis of scapular injuries X-rays are routinely taken , MSCT scanning , MRI & Nerve conduction velocity may be done.

Main parameters defining operative treatment are instability, the articular surface fragment size and the degree of displacement. However, concomitant injuries (e.g. thorax, head, extremity fractures, plexus lesion), age, occupation, level of activity and dominance, play a key role in management.

ELIGIBILITY:
Inclusion Criteria:

* 1-Fracture Pattern:

  1. All partial & complete articular Glenoid Fractures: with Non congruent articular surface; >20° deviation in angle between the glenoid and lateral scapular rim compared to the anatomical angle.
  2. All Extra articular Glenoid fractures: with >20° deviation in angle between the glenoid and lateral scapular rim compared to the anatomical angle.
  3. All Extra articular Glenoid fractures e >20° difference In GPA compared to The GPA of the normal side.
  4. Fractures e an intra-articular gap or step-off of 4 to 10 mm or more.
  5. If glenohumeral instability is present after dislocation. 2-Age: skeletally mature patients (>18-60y)

Exclusion Criteria:

* 1- Fractures e an intra-articular gap or step-off < 4 mm. 2- Timing of surgery not more than 2 weeks from the initial trauma 3- Polytraumatized patients e ISS>14. 4- Associated Neurovascular Injury. 5- Open Fractures. 6- Associated comorbidities e.g. (Uncontrolled DM, Renal impairment).

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: ALl Healthy Young Adults e out comorbidities ( DM, uncontrolled HTN,...etc)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Evaluate the role of internal fixation of glenoid fracture in healthy adults by ASES score | Baseline
  regarding functional outcome at 6 months and 1 year.

SECONDARY OUTCOMES:
Asses Fracture Union, Range of Motion Asses functional outcome by DASH score Asses Fracture Union, Range of Motion Asses functional outcome by DASH score | Baseline
  regarding functional outcome at 6 months and 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Mohamadean, Study Director — Assiut University; Galal El-Din Zaki, Study Chair — Assiut University; Mahmoud Badran, Study Director — Assiut University; Diaa El-Din Mohamed, Principal Investigator — Assiut University
Locations (1):
- ‪Diaa Mohammad‬, Asyut, Egypt

REFERENCES:
- [Background] 2.6-References : 1. Lewis Gs, Armstrong AD. glenoid spherical orientation and version. J Shoulder Elbow Surg 2011 ; 20 : 3-11. 2. Rockwood C, Matsen FAI, Wirth M, lippitt S. the shoulder. in : saunders elsevier, Philadelphia, 2009 ; 4th ed. : 333-380. 3. Van noort A. scapular fractures. in : rockwood and green's Fractures in adults. (eds. Bucholz rW, CourtBrown Cm, Heckman JD, tornetta P). Wolters Kluwer, Philadelphia, 2010 ; 7th ed : 1144-1164. 4. Jeray Kj, Cole PA. Clavicle and scapula fracture problems : functional assessment and current treatment strategies. Instr Course Lect 2011 ; 60 : 51-71. 5. Van noort A. scapular fractures. in : rockwood and green's Fractures in adults. (eds. Bucholz rW, CourtBrown Cm, Heckman JD, tornetta P). Wolters Kluwer, Philadelphia, 2010 ; 7th ed : 1144-1164. 6. Voleti PB, Namdari S, Mehta S. Fractures of the scapula. Adv Orthop. 2012;2012:1-7. doi: 10.1155/2012/903850. 7. van Oostveen, D. P. H., Temmerman, O. P. P., Burger, B. J., van Noort, A. & Robinson, M. Glenoid fractures: a review of pathology, classification, treatment and results. Acta Orthop Belg 80, 88-98 (2014). 8. Zlowodzki M, Bhandari M, Zelle BA, Kregor PJ, Cole PA. Treatment of scapula fractures: systematic review of 520 fractures in 22 case series. J Orthop Trauma. 2006;20:230-233. doi: 10.1097/00005131-200603000-00013. 9. Jaeger M, et al. The AO Foundation and Orthopaedic trauma association (AO/OTA) scapula fracture classification system: focus on glenoid fossa involvement. J Shoulder Elb Surg. 2013;22:512-520. doi: 10.1016/j.jse.2012.08.003. 10. Audige L, Kellam JF, Lambert S, et al. The AO Foundation and Orthopedic Trauma Association (AO/OTA ) scapula fracture classification system: focus in body involvement. J Shoulder Elbow surg. 2014 Feb;23 (2) :189-196. 11. Harvey E, Audige L, Herscovici D, Jr, et al. Development and validation of the new international classification for scapula fractures. J Orthop Trauma. 2012 Jun;26 (6) : 364-369. 12. Jaeger M, Lambert S, Sudkamp NP, et al. The AO Foundation and Orthopedic Trauma Association (AO/OTA ) scapula fracture classification system: focus in body involvement. J Shoulder Elbow surg. 2013 Apr; 22 (4) :512-520. 13. Bahk Ms, Kuhn j e, Galatz lM, Connor pM, Williams Gr jr. acromioclavicular and sternoclavicular injuries and clavicular, glenoid, and scapular fractures. J Bone Joint Surg Am 2009 ; 91 : 2492-2510 14. Osti M, Gohm A, Benedetto Kp. results of open reconstruction of anterior glenoid rim fractures following shoulder dislocation. Arch Orthop Trauma Surg 2009 ; 129 : 1245-1249. 15. Peter Cole, Steven R. Fractures of the Clavicle, Scapula, and Glenoid .AAOS .2014; 28:6-7.